CLINICAL TRIAL: NCT02176863
Title: A Multicenter, Prospective, Randomized, Placebo-controlled, Double-blind, Parallel-group Clinical Trial to Assess the Efficacy and Safety of Immune Globulin Intravenous (Human) Flebogamma® 5% DIF in Participants With Post-Polio Syndrome
Brief Title: Study of the Efficacy and Safety of Immune Globulin Intravenous (Human) Flebogamma® 5% Dual Inactivation and Filtration (DIF) in Participants With Post-polio Syndrome
Acronym: FORCE
Status: Terminated | Phase: Phase 2 / Phase 3 | Type: Interventional
Why Stopped: Due to Business Decision
Sponsor: Instituto Grifols, S.A. (Industry)
Responsible Party: Sponsor
Organization: Grifols Therapeutics LLC (Industry)
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: IG1104; 2013-004503-39 (EudraCT Number)
Record Dates: First submitted 2014-06-25; First posted 2014-06-27 (Estimated); Results first posted 2025-12-05 (Actual); Last update posted 2025-12-05 (Actual); Status verified 2025-11

CONDITIONS: Post-polio Syndrome
Keywords: FORCE; Post-polio syndrome; Flebogamma®; Immune Globulin Intravenous; IVIG
MeSH Terms: conditions — Postpoliomyelitis Syndrome | interventions — gamma-Globulins; Immunoglobulins, Intravenous

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Stage 1 Arm 1: 2 g/kg Flebogamma® 5% DIF (Experimental): Participants received Flebogamma® 5% DIF 2 g/kg of body weight administered via intravenous (IV) infusion over 2 consecutive days (Flebogamma® 5% DIF 1 g/kg infused on Day 1, followed by Flebogamma® 5% DIF 1 g/kg infused on Day 2) every 4 weeks for 52 weeks.
  Interventions: Biological: Flebogamma® 5% DIF
- Stage 1 Arm 2: 1 g/kg Flebogamma® 5% DIF (Experimental): Participants received Flebogamma® 5% DIF 1 g/kg of body weight administered via IV infusion on Day 1, followed by 20 mL/kg of matching placebo administered on a separate day, for a total dosing period of 2 consecutive days, every 4 weeks for 52 weeks. The order of 1 g/kg Flebogamma® 5% DIF or matching placebo was randomly determined for each participant and was the same for the participant for all infusion visits during the treatment period.
  Interventions: Biological: Flebogamma® 5% DIF; Drug: Placebo
- Stage 1 Arm 3: Placebo (Placebo Comparator): Participants received matching placebo at a total dose of 40 mL/kg of body weight administered via IV infusion over 2 consecutive days. On Day 1, a dose of 20 mL/kg of matching placebo was given, followed by the second dose of 20 mL/kg of matching placebo on Day 2, administered every 4 weeks for 52 weeks.
  Interventions: Drug: Placebo
- Stage 2 Arm 1: 1 g/kg Flebogamma® 5% DIF (Experimental): Participants received Flebogamma® 5% DIF 1 g/kg of body weight administered via IV infusion on Day 1, followed by 20 mL/kg of matching placebo administered on a separate day, for a total dosing period of 2 consecutive days, every 4 weeks for 52 weeks. The order of 1 g/kg of Flebogamma® 5% DIF or matching placebo was randomly determined for each participant and was the same for the participant for all infusion visits during the treatment period.
  Interventions: Biological: Flebogamma® 5% DIF; Drug: Placebo
- Stage 2 Arm 2: Placebo (Placebo Comparator): Participants received matching placebo at a total dose of 40 mL/kg of body weight administered via IV infusion over 2 consecutive days. On Day 1, a dose of 20 mL/kg of matching placebo was given, followed by the second dose of 20 mL/kg of matching placebo on Day 2, administered every 4 weeks for 52 weeks.
  Interventions: Drug: Placebo

INTERVENTIONS:
Biological: Flebogamma® 5% DIF — Human plasma-derived immunoglobulin
  Other Names: immune globulin intravenous (human)
  Arms: Stage 1 Arm 1: 2 g/kg Flebogamma® 5% DIF; Stage 1 Arm 2: 1 g/kg Flebogamma® 5% DIF; Stage 2 Arm 1: 1 g/kg Flebogamma® 5% DIF
Drug: Placebo — Matching placebo
  Arms: Stage 1 Arm 2: 1 g/kg Flebogamma® 5% DIF; Stage 1 Arm 3: Placebo; Stage 2 Arm 1: 1 g/kg Flebogamma® 5% DIF; Stage 2 Arm 2: Placebo

SUMMARY:
This was a multicenter, prospective, randomized, placebo-controlled, double-blind, parallel group clinical trial with adaptive dose selection in participants with post-polio syndrome (PPS).

The main purpose of this study was to select a dose of Flebogamma® 5% DIF and confirm the efficacy of the selected Flebogamma® 5% DIF dose by assessing physical performance, as measured by Two-Minute Walk Distance (2MWD) test.

The study consisted of 2 stages, with each stage consisting of a screening period (up to 4 weeks), a treatment period (52 weeks), and a follow-up period (24 weeks).

ELIGIBILITY:
Inclusion Criteria:

* Participants with Body Mass Index less than 35 kg/m^2.
* Participants who meet the clinical criteria for diagnosis of PPS as set by March-of-Dimes.
* Participants who are ambulatory or are able to walk with a cane or other aids or use a wheelchair (but they are not wheelchair-bound).
* Participants who have at least 2 newly weakened muscle groups due to PPS (as defined by medical history), with at least 1 of them in a lower extremity, and having a Medical Research Council (MRC) scale score greater than 3 at the Manual Muscle Testing (MMT) performed by the independent assessor at the Screening Visit (SV).
* Female of child-bearing potential must have a negative test for pregnancy (Human chorionic gonadotropin (HCG)-based assay).
* Female of child-bearing potential and their sexual partners have agreed to practice contraception using a method of proven reliability (i.e., hormonal methods; barrier methods; intrauterine devices methods) to prevent a pregnancy during the course of the clinical trial.
* Participants must be willing to comply with all aspects of the clinical trial protocol, including blood sampling and long-term storage of extra samples for the entire duration of the study.
* Participants who are able to walk a 2MWD of at least 50 meters at the SV and Enrollment Visit/Infusion Visit 1 (EV/IV1)
* Participants who are able to walk a consistent baseline 2 MWD, that is, the difference in 2MWD between the SV and EV/IV1 is not more than 10%.

Exclusion Criteria:

* Participants who have received human normal immune globulin treatment given by intravenous, subcutaneous, or intramuscular route within the last 3 years.
* Participants who are not ambulatory (wheelchair-bound individuals).
* Participants with poor venous access.
* Participants with intractable pain requiring narcotics or other psychotropic drugs.
* Participants with a history of anaphylactic reactions or severe reactions to any blood-derived product.
* Participants with a history of intolerance to any component of the investigational products, such as sorbitol.
* Participants receiving corticosteroids, except for those who are taking inhaled corticosteroids for asthma.
* Participants with a documented diagnosis of hyper viscosity or hypercoagulable state or thrombotic complications to polyclonal intravenous immunoglobulin (IVIG) therapy in the past.
* Participants with a history of recent (within the last year) myocardial infarction, stroke, or uncontrolled hypertension.
* Participants who suffer from congestive heart failure, embolism, or electrocardiogram changes indicative of unstable angina or atrial fibrillation.
* Participants with a history of chronic alcoholism or illicit drug abuse (addiction) in the preceding 12 months prior to the SV.
* Participants with active psychiatric illness that interferes with compliance or communication with health care personnel.
* Participants with depression with scores >30 as assessed by the Center for Epidemiologic Studies Depression (CESD) validated scale.
* Females who are pregnant or are nursing an infant child.
* Participants with any medical condition which makes clinical trial participation unadvisable or which is likely to interfere with the evaluation of the study treatment and/or the satisfactory conduct of the clinical trial according to the Investigator's judgment.
* Participants currently receiving, or have received within 3 months prior to the SV, any investigational medicinal product or device.
* Participants who are unlikely to adhere to the protocol requirements, or are likely to be uncooperative, or unable to provide a storage serum/plasma sample prior to the first investigational drug infusion.
* Participants with known selective Immune globulin A class (IgA) deficiency and serum antibodies anti-IgA.
* Participants with renal impairment (i.e., serum creatinine exceeds more than 1.5 times the upper limit of normal [ULN]) for the expected normal range for the testing laboratory).
* Participants with aspartate aminotransferase (AST) or alanine aminotransferase (ALT) levels exceeding more than 2.5 times the ULN.
* Participants with hemoglobin levels <10 g/dL, platelets levels <100,000 /mm^3, white blood cells count <3.0 k/µL, and erythrocyte sedimentation rate >50 mm/h or twice above normal.
* Participants with known seropositive to Hepatitis C virus (HCV), Human immunodeficiency virus-1 (HIV-1) and/or Human immunodeficiency virus-2 (HIV-2).
* Participants with a history of intolerance to fructose.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 191 (Actual)
Dates: Start 2014-09-23 (Actual); Primary Completion 2022-11-24 (Actual); Study Completion 2022-11-24 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Marinos Dalakas, MD, Principal Investigator — Coordinating Investigator
Locations (21):
- United States (4):
  - Washington University, St Louis, Missouri
  - SUNY Upstate Medical University, Syracuse, New York
  - Thomas Jefferson University Hospital, Philadelphia, Pennsylvania
  - Medical College of Wisconsin, Milwaukee, Wisconsin
- Montreal Neurological Institute Clinical Research Unit, McGill University, Montreal, Quebec, Canada
- Thomayerova nemocnice, Klinicko-farmakologická jednotka, Prague, Czechia
- Denmark (2):
  - Aarhus Universitets Hospital-Neurologisk Forskning, Aarhus N
  - Rigshospitalet, København Ø
- Germany (5):
  - Charité Campus Mitte, Berlin
  - Hannover Medical School, Hanover
  - Universitätsklinikum Jena, Jena
  - Klinik für konservative Orthopädie und des Poliozentrums, Koblenz
  - Westfälische Wilhelms-Universität Münster, Münster
- Azienda Ospedaliera Universitaria Integrata Verona (Ospedale Borgo Roma), Verona, Italy
- Academisch Medisch Centrum Amsterdam UMC, Locatie AMC, Amsterdam, Netherlands
- Poland (4):
  - MedTrials, Krakow
  - Samodzielny Publiczny Szpital Kliniczny Nr 4 w Lublinie, Lublin
  - Clinical Research Center Sp. z o.o., Poznan
  - Samodzielny Publiczny Centralny Szpital Kliniczny, Warsaw
- Spain (2):
  - Institut Guttman, Badalona
  - Hospital Universitari Vall d'Hebron, Barcelona

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants took part in the study from 23 September 2014 to 24 November 2022.
Pre-assignment Details: A total of 238 participants were screened, out of which 191 participants were randomized in the study. Participants with post-polio syndrome (PPS) were randomized to receive Flebogamma® 5% DIF or placebo during Stage 1 or 2 of the study. During Stage 1, 161 participants were screened, of which 126 participants were randomized in the study. During Stage 2, 77 participants were screened, of which 65 participants were randomized in the study.
Period: Overall Study
Arm/Group | Stage 1 Arm 1: 2 g/kg Flebogamma® 5% DIF | Stage 1 Arm 2: 1 g/kg Flebogamma® 5% DIF | Stage 1 Arm 3: Placebo | Stage 2 Arm 1: 1 g/kg Flebogamma® 5% DIF | Stage 2 Arm 2: Placebo
Started | 42 | 42 | 42 | 33 | 32
Completed | 25 | 34 | 33 | 26 | 26
Not Completed | 17 | 8 | 9 | 7 | 6
Not completed — Physician Decision | 1 | 0 | 0 | 0 | 0
Not completed — Adverse Event | 10 | 4 | 4 | 1 | 1
Not completed — Protocol Violation | 2 | 0 | 1 | 1 | 0
Not completed — Withdrawal by Subject | 4 | 2 | 2 | 3 | 4
Not completed — Reason not specified | 0 | 1 | 1 | 2 | 1
Not completed — Lost to Follow-up | 0 | 1 | 1 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included all participants who were randomized.
Groups:
- Total: Total of all reporting groups
Arm/Group | Stage 1 Arm 1: 2 g/kg Flebogamma® 5% DIF | Stage 1 Arm 2: 1 g/kg Flebogamma® 5% DIF | Stage 1 Arm 3: Placebo | Stage 2 Arm 1: 1 g/kg Flebogamma® 5% DIF | Stage 2 Arm 2: Placebo | Total
Number analyzed (Participants) | 42 | 42 | 42 | 33 | 32 | 191
Age, Continuous [Mean (Standard Deviation); unit: years] | 63.3 (6.24) | 62.3 (6.88) | 62.2 (7.22) | 65.1 (7.00) | 63.9 (6.26) | 63.2 (6.76)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 23 | 21 | 27 | 22 | 22 | 115
  Male | 19 | 21 | 15 | 11 | 10 | 76
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 3 | 6 | 6 | 4 | 1 | 20
  Not Hispanic or Latino | 39 | 36 | 36 | 29 | 31 | 171
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0 | 0
  Asian | 2 | 2 | 1 | 1 | 0 | 6
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0 | 0
  Black or African American | 0 | 0 | 1 | 1 | 0 | 2
  White | 40 | 40 | 40 | 31 | 31 | 182
  More than one race | 0 | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 1 | 1

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Physical Performance Assessed by Two-Minute Walk Distance (2MWD) Test
Description: The 2MWD was used to assess physical performance by measuring the distance that a participant can quickly walk at a self-preferred speed on an indoor flat, hard surface 30 m (100-ft) hallway in a period of 2 minutes. A positive change from baseline indicates improvement (i.e. a patient can walk farther). Increase in distance walked (in meters) indicates improvement.
Time Frame: Baseline to Week 52
Population: ITT population included all participants who were randomized.
Measure: Mean (Standard Deviation); unit: meters (m)
Arm/Group | Stage 1 Arm 1: 2 g/kg Flebogamma® 5% DIF | Stage 1 Arm 2: 1 g/kg Flebogamma® 5% DIF | Stage 1 Arm 3: Placebo | Stage 2 Arm 1: 1 g/kg Flebogamma® 5% DIF | Stage 2 Arm 2: Placebo
Number analyzed (Participants) | 42 | 42 | 42 | 33 | 32
meters (m)
  Baseline | 109.03 (30.564) | 112.55 (27.987) | 105.86 (31.942) | 101.18 (22.588) | 107.10 (30.167)
  Change from Baseline at Week 52 | 7.50 (14.666) | 10.89 (19.067) | 3.17 (11.080) | 11.31 (12.108) | 5.65 (10.388)
Statistical Analysis 1: Comparison: Stage 1 Arm 2: 1 g/kg Flebogamma® 5% DIF vs Stage 1 Arm 3: Placebo vs Stage 2 Arm 1: 1 g/kg Flebogamma® 5% DIF vs Stage 2 Arm 2: Placebo; Test type: Superiority; p = 0.0469, Posch and Bauer Method — The overall adjusted p-value for the selected dose of Flebogamma® 5% DIF vs placebo was calculated from the p-values of both Stage 1 and Stage 2 by Posch & Bauer for testing the equality of means between the selected dose and placebo

2. Secondary Outcome: Change From Baseline in Pain Using Visual Analogue Scale (VAS) of Pain
Description: VAS is a participant self-reported pain scale used to evaluate the pain level in a 24 hours period. The scale consists of a 100 millimeters (mm) scale where 100 mm stands for the worst imaginable pain and zero stands for no pain. Higher scores indicate severe pain. A negative change from baseline indicates improvement. LS mean and 95% (CI) were based on MMRM method.
Time Frame: Baseline to Week 52
Population: ITT population included all participants who were randomized. As pre-specified in SAP, the analyses was performed over the two stages combined, using the placebo and selected dose of Flebogamma® 5% DIF treatment groups.
Measure: Least Squares Mean (95% Confidence Interval); unit: millimeter (mm)
Groups:
- Flebogamma® 5% DIF 1 g/kg: Participants received Flebogamma® 5% DIF 1 g/kg of body weight administered via IV infusion on Day 1 followed by 20 mL/kg of matching placebo administered on a separate day, for a total dosing period of 2 consecutive days every 4 weeks for 52 weeks during Stage 1 and then every 4 weeks for 52 weeks during Stage 2 of the study. The order of 1 g/kg of Flebogamma® 5% DIF was randomly determined for each participant and was the same for the participant for all infusion visits during the treatment period.
- Placebo: Participants received matching placebo at a total dose of 40 mL/kg of body weight administered via IV infusion over 2 consecutive days. On Day 1, a dose of 20 mL/kg of matching placebo was given, followed by the second dose of 20 mL/kg of matching placebo on Day 2, administered every 4 weeks for 52 weeks during Stage 1 and then every 4 weeks for 52 weeks during Stage 2 of the study.
Arm/Group | Flebogamma® 5% DIF 1 g/kg | Placebo
Number analyzed (Participants) | 75 | 74
millimeter (mm) | -3.2 [-10.4 to 4.1] | -2.6 [-9.9 to 4.6]
Statistical Analysis 1: Comparison: Flebogamma® 5% DIF 1 g/kg vs Placebo; Test type: Superiority; p = 0.8897, Mixed-effect Model Repeated Measures — MMRM include change from baseline in VAS as dependent variable;treatment,protocol-specified visit,treatment-by-visit interaction,main part affected(fixed effect);baseline as covariate & measures within-participants at each visit(repeated measure); LS Mean Difference = -0.5, 95% CI 2-sided [-7.7 to 6.7], Standard Error of Mean 3.65

3. Secondary Outcome: Change From Baseline in Health-Related Quality of Life (HRQoL) Assessed by Medical Outcomes Study 36-Item Short-Form Health Survey (SF-36) Physical Component Summary (PCS)
Description: HRQoL SF-36 is participant self-reported survey.It yields 8-scale profile of functional health and well-being as well as physical and mental health summary measures. It consists of the subscales:physical functioning,limitations due to physical health,body pain,general health,vitality,social functioning,emotional problems, and mental health. Each domain score ranges from 0(worst) to 100(best),higher scores reflect better functional status.PCS is a subscale score & give broader metric of physical HRQoL.PCS score ranges from 0 to 100 and is computed such that mean score of 50 corresponds to the general US population.Based on norm-based scoring,scores above 50 is better-than-average health & below 50 is below-average health.Higher scores represents better physical health.Positive change from baseline indicates improvement.LS mean and 95% CI were based on MMRM.
Time Frame: Baseline to Week 52
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: Score on a scale
Arm/Group | Flebogamma® 5% DIF 1 g/kg | Placebo
Number analyzed (Participants) | 75 | 74
Score on a scale | 4.78 [1.9 to 7.6] | 2.79 [-0.1 to 5.7]
Statistical Analysis 1: Comparison: Flebogamma® 5% DIF 1 g/kg vs Placebo; Test type: Superiority; p = 0.1615, Mixed-effect Model Repeated Measures — MMRM include change from baseline in SF-36PCS as dependent variable;treatment protocol-specified visit,treatment-by-visit interaction,main part affected(fixed effect);baseline measure as covariate & within-participant at each visit(repeated measure); LS Mean Difference = 1.98, 95% CI 2-sided [-0.8 to 4.8], Standard Error of Mean 1.410

4. Secondary Outcome: Change From Baseline in Endurance Assessed by Six-Minute Walk Distance (6MWD) Test
Description: The 6MWD was used to assess physical performance by measuring the distance that a patient can quickly walk at maximal speed on a flat, hard surface 30 m (100-ft) hallway in a period of 6 minutes. A positive change from baseline indicates improvement (i.e., a patient can walk farther). Increase from baseline in distance walked (in meters) indicated improvement. LS mean and 95% CI were based on MMRM method.
Time Frame: Baseline to Week 52
Population: as for outcome 2
Measure: Least Squares Mean (95% Confidence Interval); unit: meters (m)
Arm/Group | Flebogamma® 5% DIF 1 g/kg | Placebo
Number analyzed (Participants) | 75 | 74
meters (m) | 29.16 [7.54 to 50.78] | 13.36 [-8.22 to 34.95]
Statistical Analysis 1: Comparison: Flebogamma® 5% DIF 1 g/kg vs Placebo; Test type: Superiority; p = 0.1205, Mixed-effect Model Repeated Measures — MMRM include change from baseline in 6MWD as dependent variable;treatment,protocol-specified visit,treatment-by-visit interaction,main part affected(fixed effect);baseline as covariate & measures within-participants at each visit(repeated measure); LS Mean Difference = 15.80, 95% CI 2-sided [-4.19 to 35.79], Standard Error of Mean 10.112

ADVERSE EVENTS:
Time Frame: From the start of study drug administration through 4 weeks after last study treatment (Up to Week 56)
Description: The Safety population included all participants who received at least 1 infusion of investigational product (Flebogamma® 5% DIF or placebo). As pre-specified in the SAP, the combined safety data from both Stage 1 and Stage 2 together was summarized by treatment arm. Safety analyses was performed according to the actual treatment received. Only On Treatment Treatment-Emergent Adverse Events have been reported.
Groups:
- Flebogamma® 5% DIF 2 g/kg: Participants received Flebogamma® 5% DIF 2 g/kg of body weight administered via intravenous (IV) infusion over 2 consecutive days (Flebogamma® 5% DIF 1 g/kg infused on Day 1, followed by Flebogamma® 5% DIF 1 g/kg infused on Day 2) every 4 weeks for 52 weeks.
Arm/Group | Flebogamma® 5% DIF 2 g/kg | Flebogamma® 5% DIF 1 g/kg | Placebo
All-Cause Mortality (participants affected / at risk) | 0/42 | 0/75 | 0/74
Serious Adverse Events (participants affected / at risk) | 3/42 | 7/75 | 9/74
Other Adverse Events (participants affected / at risk) | 36/42 | 71/75 | 60/74
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Flebogamma® 5% DIF 2 g/kg (N=42) | Flebogamma® 5% DIF 1 g/kg (N=75) | Placebo (N=74)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0
Hypertension (Vascular disorders) | 0 | 0 | 2
Miscarriage of partner (Social circumstances) | 0 | 0 | 1
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0
Diagnostic procedure (Investigations) | 0 | 1 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1
Bone fissure (Injury, poisoning and procedural complications) | 0 | 0 | 1
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0
Myocardial infarction (Cardiac disorders) | 1 | 0 | 0
Meningism (Nervous system disorders) | 0 | 1 | 0
Syncope (Nervous system disorders) | 0 | 0 | 1
Vertigo positional (Ear and labyrinth disorders) | 0 | 1 | 0
Food poisoning (Gastrointestinal disorders) | 0 | 0 | 1
Pancreatitis chronic (Gastrointestinal disorders) | 0 | 0 | 1
Acute kidney injury (Renal and urinary disorders) | 0 | 0 | 1
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0
Herpes zoster (Infections and infestations) | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 0 | 2
Prostate infection (Infections and infestations) | 0 | 1 | 0
Pyelonephritis (Infections and infestations) | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Flebogamma® 5% DIF 2 g/kg (N=42) | Flebogamma® 5% DIF 1 g/kg (N=75) | Placebo (N=74)
Vertigo (Ear and labyrinth disorders) | 2 | 3 | 4
Diarrhoea (Gastrointestinal disorders) | 0 | 7 | 8
Nausea (Gastrointestinal disorders) | 11 | 13 | 4
Vomiting (Gastrointestinal disorders) | 6 | 5 | 3
Chills (General disorders) | 8 | 15 | 2
Fatigue (General disorders) | 14 | 22 | 20
Influenza like illness (General disorders) | 0 | 10 | 3
Infusion site swelling (General disorders) | 2 | 2 | 4
Non-cardiac chest pain (General disorders) | 2 | 4 | 1
Oedema peripheral (General disorders) | 2 | 3 | 8
Pain (General disorders) | 3 | 5 | 1
Pyrexia (General disorders) | 8 | 13 | 1
Cystitis (Infections and infestations) | 1 | 2 | 4
Influenza (Infections and infestations) | 4 | 9 | 2
Nasopharyngitis (Infections and infestations) | 4 | 8 | 11
Contusion (Injury, poisoning and procedural complications) | 1 | 3 | 4
Fall (Injury, poisoning and procedural complications) | 2 | 5 | 8
Blood pressure increased (Investigations) | 0 | 8 | 0
Fibrin D dimer increased (Investigations) | 3 | 5 | 5
Arthralgia (Musculoskeletal and connective tissue disorders) | 8 | 12 | 12
Back pain (Musculoskeletal and connective tissue disorders) | 5 | 8 | 6
Muscular weakness (Musculoskeletal and connective tissue disorders) | 1 | 2 | 4
Myalgia (Musculoskeletal and connective tissue disorders) | 6 | 10 | 3
Neck pain (Musculoskeletal and connective tissue disorders) | 0 | 4 | 2
Pain in extremity (Musculoskeletal and connective tissue disorders) | 3 | 10 | 5
Dizziness (Nervous system disorders) | 3 | 4 | 13
Headache (Nervous system disorders) | 27 | 39 | 23
Hypoaesthesia (Nervous system disorders) | 1 | 4 | 3
Migraine (Nervous system disorders) | 2 | 5 | 1
Paraesthesia (Nervous system disorders) | 0 | 5 | 4
Device dislocation (Product Issues) | 3 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 4 | 0
Cough (Respiratory, thoracic and mediastinal disorders) | 4 | 3 | 1
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 4 | 1 | 3
Oropharyngeal pain (Respiratory, thoracic and mediastinal disorders) | 0 | 4 | 2
Dry skin (Skin and subcutaneous tissue disorders) | 1 | 4 | 0
Eczema (Skin and subcutaneous tissue disorders) | 0 | 4 | 1
Erythema (Skin and subcutaneous tissue disorders) | 2 | 4 | 1
Pruritus (Skin and subcutaneous tissue disorders) | 2 | 7 | 3
Rash (Skin and subcutaneous tissue disorders) | 1 | 11 | 0
Hypertension (Vascular disorders) | 7 | 12 | 8
Phlebitis (Vascular disorders) | 3 | 3 | 0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Site may publish results from the Study, after providing Sponsor 30 days' notice prior to submitting a manuscript or other materials related to the Study to any outside party. At the Sponsors' request, the Site will remove any Confidential Information (other than Study results), and the Site will upon Sponsors' request, delay publication or presentation for a period of up to 120 days to allow the Sponsor to protect its interests in any Sponsor Inventions.

DOCUMENTS (2):
  • Study Protocol (2022-03-07): https://cdn.clinicaltrials.gov/large-docs/63/NCT02176863/Prot_000.pdf
  • Statistical Analysis Plan (2023-08-28): https://cdn.clinicaltrials.gov/large-docs/63/NCT02176863/SAP_001.pdf